

## Direzione Ricerca, Innovazione e Internazionalizzazione

## Prot. n.\*

n. e data della registrazione di protocollo riportati nei metadati del sistema di protocollo informatico Titulus

> Al Prof. Ilario Ferrocino Dipartimento di Scienze Agrarie, Forestali ed Alimentari Largo Braccini, 2 Grugliasco (Torino)

Oggetto: Parere progetto

Si comunica che in data 17 giugno 2024 il Comitato di Bioetica d'Ateneo ha espresso parere favorevole per il progetto di ricerca dal titolo: "ALIMENTI FUNZIONALIZZATI ARRICCHITI CON PROTEINE DI GRILLO E PROTEINE DI ORIGINE VEGETALE (NOODLE)".

Cordiali saluti

(Segreteria Comitato di Bioetica d'Ateneo)

Cesarina Marretta



## MODULO DI CONSENSO INFORMATO

## dichiaro

- di non avere patologie acute o croniche che richiedano specifici trattamenti farmacologici o restrizioni dietetiche e di non avere allergia o intolleranze all'alimento da testare:
- ✓ di partecipare volontariamente allo studio;
- ✓ di aver ricevuto dal Prof. Ilario Ferrocino o dai suoi collaboratori esaurienti spiegazioni in merito alla richiesta di partecipazione alla ricerca, in particolare sulle finalità e procedure;
- di aver avuto a disposizione tempo sufficiente per poter leggere attentamente, comprendere ed eventualmente farmi spiegare quanto contenuto nella scheda informativa allegata e da me sottoscritta per presa visione, e che conferma quanto mi è stato spiegato a voce, in particolare che la sperimentazione sarà condotta nel rispetto dei codici etici internazionali;
- di aver avuto la possibilità di porre domande e di aver avuto risposte soddisfacenti su tutta la sperimentazione ed in particolare sulle possibili alternative diagnostiche e terapeutiche e sulle conseguenze della mancata esecuzione della procedura proposta;
- ✓ di essere stato informato sui possibili rischi o disagi ragionevolmente prevedibili;
- ✓ di acconsentire che il medico responsabile informi il mio medico di famiglia;





- ✓ di acconsentire che i monitor, audit, autorità regolatorie nazionali ed estere abbiano accesso diretto alla mia documentazione clinica ai fini di monitoraggio e verifica;
- di essere consapevole che la partecipazione è volontaria, con l'assicurazione che il rifiuto a partecipare non influirà nel ricevere il trattamento più idoneo;
- che potrò ritirarmi dalla sperimentazione già iniziata in qualsiasi momento, senza conseguenze negative nel ricevere il trattamento più idoneo e senza l'obbligo da parte mia di motivarne la decisione, a meno che la stessa non derivi dalla comparsa di disturbi o effetti indesiderati e/o non previsti, nel qual caso mi impegno fin da ora a comunicarne tempestivamente agli sperimentatori natura ed entità;
- ✓ che i dati clinici resteranno strettamente riservati e saranno utilizzati con le finalità indicate nello studio (GDPR, Reg.UE n. 2016/679, D. Lgs. n. 101/2018 e come da Linee Guida del Garante per il trattamento dei dati personali nell'ambito delle sperimentazioni cliniche di medicinali (G.U. 190 del 14/08/2008) e come da ogni altra prescrizione/autorizzazione del Garante stesso);
- ✓ che sarò informato di eventuali nuovi dati che possano influenzare i rischi o i benefici, oppure di variazioni di protocollo che possano influenzarli;
- ✓ di essere stato informato che è mio diritto avere accesso alla documentazione che mi riguarda e alla valutazione espressa dal Comitato Etico cui potrò rivolgermi se lo terrò opportuno
- ✓ che una copia del consenso informato e della documentazione di cui ho preso visione rimarrà in mio possesso; che per ogni problema o per eventuali ulteriori informazioni potrò rivolgermi al Medico Sperimentatore:

Prof. Ilario Ferrocino DISAFA - Microbiology and food technology sector. Università degli Studi di Torino.

Recapito telefonico: 011-6708847

e-mail: studiomicrobiota2020@gmail.com



| ACCONSENTO |
|---|
| LIBERAMENTE, SPONTANEAMENTE E IN PIENA COSCIENZA ALLO STUDIO PROPOSTOMI |
| Dichiaro inoltre di essere a conoscenza della possibilità di revocare il presente consenso in qualsiasi momento prima dell'avvio della sperimentazione. DataOra inizio colloquioOra fine |
| colloquio |
| Eventuali testimoni presenti (nome, cognome, firma): |
| Firma del partecipante |
| Firma dello sperimentatore |
| oppure |
| NON ACCONSENTO |
| LIBERAMENTE, SPONTANEAMENTE E IN PIENA COSCIENZA ALLO STUDIO PROPOSTOMI DataOra inizio colloquioOra fine |
| colloquio |
| Eventuali testimoni presenti (nome, cognome, firma): |
| Firma del partecipante |
| Firma dello sperimentatore |
| DICHIARAZIONE DELL'INCARICATO DELLA SPERIMENTAZIONE. |
| Io sottoscritto, confermo ed attesto, in |
| modo consensuale alla sottoscrizione della persona consenziente, che la stessa a mio |
| avviso, ha interamente compreso tutto quanto sopra esposto, punto per punto. |
| Data |



| luogo ed o | ra | <br> | <br> | <br> | <br> | <br> | <br> | <br> |
|------------|----|------|------|------|------|------|------|------|
| In fede | | <br> | <br> | <br> | <br> | <br> | <br> | <br> |